CLINICAL TRIAL: NCT01433172
Title: A Randomized Phase I/II Trial Using a GM-CSF-Producing and CD40L-Expressing Bystander Cell Line (GM.CD40L) Vaccine in Combination With CCL21 for Patients With Stage IV Adenocarcinoma of the Lung
Brief Title: Combination Immunotherapy of GM.CD40L Vaccine With CCL21 in Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bankhead-Coley Florida Biomedical Research Program (Unknown); James and Esther King Biomedical Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16439
Record Dates: First submitted 2011-09-12; First posted 2011-09-13 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Lung Cancer; Adenocarcinoma
Keywords: stage IV; adenocarcinoma; vaccine therapy; immunology; tumor vaccine; colony stimulating factor(CSF); granulocyte-macrophage colony-stimulating factor (GM-CSF); CC chemokine ligand 21 (CCL21); Chemokine [C-C motif] ligand 21 (CCL21); human leukocyte antigen serotype (HLA)
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma | interventions — Chemokines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase I Vaccinations (Experimental): Participants enrolled in the Phase I trial will receive GM.CD40L.CCL21 vaccinations on 3 occasions, at 2 week intervals. Note for the phase I portion: the use of steroid medication is to be avoided for 4 weeks prior to the initiation of vaccine therapy and during the vaccine treatment period.
  Interventions: Biological: Phase I - GM.CD40L.CCL21 Vaccinations
- Phase II Arm A Vaccinations (Active Comparator): Arm A participants will receive GM.CD40L cells vaccinations on 3 occasions, at 2 week intervals. Note on either Arms A and B: the use of steroid medication is to be avoided for 4 weeks before to the initiation of vaccine therapy and during the vaccine treatment period.
  Interventions: Biological: Phase II - GM.CD40L cells Vaccinations
- Phase II Arm B Vaccinations (Active Comparator): Arm B participants will receive GM.CD40L.CCL21 vaccinations on 3 occasions, at 2 week intervals. Note on either Arms A and B: the use of steroid medication is to be avoided for 4 weeks before to the initiation of vaccine therapy and during the vaccine treatment period.
  Interventions: Biological: Phase II - GM.CD40L.CCL21 Vaccinations

INTERVENTIONS:
Biological: Phase I - GM.CD40L.CCL21 Vaccinations — This is a dual-agent, Phase I study with an expansion of each group at the recommended Phase II dose. Participants are entered in cohorts of 3 at the first dose level. Doses are not escalated over the course of treatment of an individual patient.
  Phase I: Participants receive the GM.CD40L.CCL21 vaccine in a standard 3+3 design.
  Other Names: chemokine
  Arms: Phase I Vaccinations
Biological: Phase II - GM.CD40L cells Vaccinations — Patients randomized to Arm A will receive vaccinations on 3 occasions, at 2 week intervals. 7.5 X 10^6 irradiated H1944 tumor cells, 7.5 X 10^6 irradiated H2122 cells, and containing 15 X 10^6 GM.CD40L cells (1.1 mL) will be injected intradermally into 4 separate sites (0.25 ml injected at each site), in bilateral proximal upper and lower extremities (in the regions of the axillary and inguinal nodal basins). Patients will be restaged approximately 2 weeks after vaccine 3. If patients show no sign of disease progression, patients will then be vaccinated at 4-week intervals.
  Other Names: MHC-negative cell line
  Arms: Phase II Arm A Vaccinations
Biological: Phase II - GM.CD40L.CCL21 Vaccinations — This is a dual-agent, Phase I study with an expansion of each group at the recommended Phase II dose. Participants are entered in cohorts of 3 at the first dose level. Doses are not escalated over the course of treatment of an individual patient.
  Phase II: Participants are randomized to one of the 2 arms (ratio 1:1): GM.CD40L versus GM.CD40L.CCL21. Patients in Arm B will receive vaccines at the same dose and schedule as described for patients in Arm A. In addition, their vaccine will include H1944 cells expressing CCL21. Note for patients on Arms A and B: the use of steroid medication is to be avoided for 4 weeks before to the initiation of vaccine therapy and during the vaccine treatment period.
  Other Names: chemokine
  Arms: Phase II Arm B Vaccinations

SUMMARY:
The purpose of this study is to find out what effects (good and bad) a tumor vaccine used in combination with GM.CD40L and CCL21 have on the patient and their cancer. We also want to find out if the vaccine and the drugs can boost the immune system of these patients and how their immune system reacts, both before and after the vaccine treatment.

DETAILED DESCRIPTION:
The vaccine will be made by mixing two kinds of cells: 1) some lung cancer cells, which have been grown in the lab, and 2) experimental "bystander (present but not taking part in the immune response)" cells. All the cells in the vaccine will be treated with high-dose X-rays to make sure that none of them grow and cause more cancer. The bystander cells are human cells that have been genetically changed to express GM-CSF and CD40L. These are called "GM.CD40L". (That is the original cells, called K562, with the genes for human GM-CSF and CD40L inserted into them). These changes are designed to help boost the participants' immune system to better fight the cancer in their body. GM-CSF is a hormone that is known to stimulate bone marrow to make more white blood cells.

CCL21 is a chemokine (protein) that helps to recruit T cells (a type of white blood cell that helps to protect the body from infections) and leads to hyper-responsive T cells. This leads to heightened immune responses when T cells are exposed to both CCL21 and antigen (a substance that when introduced into the body lead to production of an antibody)-presenting cells (A cell that can "present" antigen in a form that T cells can recognize it ). The induction of a strong cell-mediated immune response is the type of immunity expected to be most involved in controlling cancer cell growth. A randomized trial of a vaccine consisting of the GM.CD40L bystander cells and an equivalent number of allogeneic (taken from different individuals) tumor cells plus or minus CCL21 is proposed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic adenocarcinoma of the lung
* Patients must have received and completed first line therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, or 1
* No external beam radiation therapy within 2 weeks of first vaccine administration
* No stereotactic radiation therapy within 3 days of first vaccine
* No targeted therapy within 2 weeks of first vaccine administration
* No immunomodulatory therapy within 2 weeks of first vaccine administration
* No chemotherapy within 4 weeks of first vaccine administration
* During Screening period, no steroid therapy within 4 weeks of first vaccine administration
* Patient's written informed consent
* Adequate organ function (measured within a week of beginning treatment):

  * White blood count (WBC) > 3,000/mm³ and absolute neutrophil count (ANC) >/= 1500/mm³
  * Platelets > 100,000/mm³
  * Hematocrit > 25%
  * Bilirubin < 2.0 mg/dL
  * Creatinine < 2.0 mg/dL, or creatinine clearance > 60 mL/min
* Patients will be tested for HLA-A0201 as determined by flow cytometry followed by molecular analysis of a peripheral blood specimen; however this result will not be an inclusion criterion.
* Measurable metastatic tumor as defined by standard Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Lesions must be accurately measured in at least one dimension with the longest diameter ≥20 mm. With spiral computed tomography (CT) scan, lesion must be ≥10 mm in at least one dimension.

Exclusion Criteria:

* Symptomatic brain metastasis or Uncontrolled central nervous system (CNS) metastasis will not be permitted.
* Any acute medical problems requiring active intervention
* Current corticosteroid (other than replacement doses in patients who are hypo-adrenal) or other immunosuppressive therapy
* Any other pre-existing immunodeficiency condition (including known human immunodeficiency virus [HIV] infection)
* Any known pre-existing autoimmune disorder
* History of a second malignancy within the previous 2 years (except non-melanoma skin cancer and cervical in-situ)
* Patients who have had major surgery without full recovery or major surgery within three weeks of the start of vaccine treatment
* Pregnant or lactating women: Patients in reproductive age must agree to use contraceptive methods for the duration of the study (*A pregnancy test will be obtained before treatment).
* Eastern Cooperative Oncology Group (ECOG) performance status of 2, 3, or 4
* Patients with other significant diseases or disorders that, in the Investigator's opinion, would exclude them from the study.
* Patients who at the discretion of the investigator are deemed to have rapidly progressive disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-03-26 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2019-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jhanelle Gray, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Moffitt Cancer Center between April 2012 and June 2015.
Pre-assignment Details: Three participants were enrolled in the Phase I portion of the study, followed by seventy participants enrolled in the Randomized Phase II portion of the study.
Groups:
- Phase I GM.CD40L.CCL21 Vaccinations: Participants enrolled in the Phase I trial will receive GM.CD40L.CCL21 vaccinations on 3 occasions, at 2 week intervals. Note for the phase I portion: the use of steroid medication is to be avoided for 4 weeks prior to the initiation of vaccine therapy and during the vaccine treatment period.
- Phase II Arm A GM.CD40L Cells Vaccinations: Phase II Arm A: Participants will receive GM.CD40L cells vaccinations on 3 occasions, at 2 week intervals. Note on either Arms A and B: the use of steroid medication is to be avoided for 4 weeks before to the initiation of vaccine therapy and during the vaccine treatment period.
- Phase II Arm B GM.CD40L.CCL21 Vaccinations: Phase II Arm B: Participants will receive GM.CD40L.CCL21 vaccinations on 3 occasions, at 2 week intervals. Note on either Arms A and B: the use of steroid medication is to be avoided for 4 weeks before to the initiation of vaccine therapy and during the vaccine treatment period.
Period: Overall Study
Arm/Group | Phase I GM.CD40L.CCL21 Vaccinations | Phase II Arm A GM.CD40L Cells Vaccinations | Phase II Arm B GM.CD40L.CCL21 Vaccinations
Started | 3 | 37 | 33
Completed | 3 | 34 | 32
Not Completed | 0 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Disease Progression | 0 | 0 | 1
Not completed — Death | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All participants.
Groups:
- Phase I Vaccinations: Participants enrolled in the Phase I trial will receive GM.CD40L.CCL21 vaccinations on 3 occasions, at 2 week intervals.
- Phase II Arm A Vaccinations: Arm A participants will receive GM.CD40L cells vaccinations on 3 occasions, at 2 week intervals.
- Phase II Arm B Vaccinations: Arm B participants will receive GM.CD40L.CCL21 vaccinations on 3 occasions, at 2 week intervals.
- Total: Total of all reporting groups
Arm/Group | Phase I Vaccinations | Phase II Arm A Vaccinations | Phase II Arm B Vaccinations | Total
Number analyzed (Participants) | 3 | 37 | 33 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 16 | 10 | 27
  >=65 years | 2 | 21 | 23 | 46
Age, Continuous [Median (Full Range); unit: years] | 68 [58 to 78] | 62 [38 to 86] | 65 [48 to 82] | 62 [38 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 19 | 19 | 38
  Male | 3 | 18 | 14 | 35
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 37 | 33 | 73

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Recommend Phase II Dose (RPDII)
Description: Highest dose level of GMCD40L vaccine in combination with CCL21 that induced dose limiting toxicity (DLT) in fewer than 33% of patients. DLT: Intervention-specific acute toxicity; i.e., occurrence within 28 days of drug administration, according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), V 4: 1.) that precludes further dose escalation. Participants are entered in cohorts of 3 at the first dose level. Doses are not escalated over the course of treatment of an individual patient. If 2 or more patients experience toxicity in dose level 1 (30X10^6 cells per injection), dose de-escalation will occur. Dose level -1 will be defined by 10 % reduction of cells administered from dose level 1 and follow the same rules. It is not feasible to escalate the dose of the vaccine beyond 30X10^6 cells per injection; therefore the Maximum Tolerated Dose (MTD) may not be reached in this study. In that case, the highest dose level will be used in the phase II component.
Time Frame: Up to 6 Months
Population: All Phase I Participants
Measure: Number; unit: Recommend Phase II Dose Level
Groups:
- Phase I GM.CD40L.CCL21 Vaccinations: Participants enrolled in the Phase I trial will receive GM.CD40L.CCL21 vaccinations on 3 occasions, at 2 week intervals.
Arm/Group | Phase I GM.CD40L.CCL21 Vaccinations
Number analyzed (Participants) | 3
Recommend Phase II Dose Level | 1

2. Primary Outcome: Phase II: Progression Free Survival (PFS)
Description: PFS is measured as the time from start of treatment to progression or death. 6 month progression free survival will be estimated from available clinical and radiographic assessments and RECIST 1.1 will be used to make tumor measurements. Progressive Disease (PD) = 20% increase in the sum of the longest diameter of target lesions.
Time Frame: Up to 6 Months
Population: A Phase II participants evaluable at time of analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase II Arm A GM.CD40L Cells Vaccinations: Arm A participants will receive GM.CD40L cells vaccinations on 3 occasions, at 2 week intervals.
- Phase II Arm B GM.CD40L.CCL21 Vaccinations: Arm B participants will receive GM.CD40L.CCL21 vaccinations on 3 occasions, at 2 week intervals.
Arm/Group | Phase II Arm A GM.CD40L Cells Vaccinations | Phase II Arm B GM.CD40L.CCL21 Vaccinations
Number analyzed (Participants) | 33 | 32
months | 2.4 [1.6 to 4.4] | 3.1 [1.6 to 4.4]

3. Secondary Outcome: Response Rate
Description: Response according to Response Evaluation in Solid Tumors (RECIST) 1.1. Complete Response (CR): Complete disappearance of all measurable and non-measurable disease; No new lesions. Partial Response (PR): Applies only to patients with at least one measurable lesion; Greater than or equal to 30% decrease under baseline of the sum of longest diameters of all target measurable lesions. Progressive Disease (PD): 20% or greater increase in the sum of longest diameters of target measurable lesions over smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline. Unequivocal progression of non-measurable disease in the opinion of the treating physician (an explanation must be provided). Appearance of any new lesion/site. Stable Disease (SD): Does not qualify for CR, PR, Progression or Symptomatic Deterioration; All target measurable lesions must be assessed using the same techniques as baseline.
Time Frame: Up to 12 Months
Population: All Phase II participants
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II Arm A GM.CD40L Cells Vaccinations | Phase II Arm B GM.CD40L.CCL21 Vaccinations
Number analyzed (Participants) | 37 | 33
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 0
  Progressive Disease | 19 | 20
  Stable Disease | 18 | 12

ADVERSE EVENTS:
Time Frame: 3 years, 8 months
Description: All Serious Adverse Events and Other (not including Serious) Adverse Events are listed, regardless of causality. All SAEs were either not related or unlikely to be related to study vaccines.
Groups:
- Phase II Arm A GM.CD40L Vaccinations: Arm A participants will receive GM.CD40L cells vaccinations on 3 occasions, at 2 week intervals.
Arm/Group | Phase I GM.CD40L.CCL21 Vaccinations | Phase II Arm A GM.CD40L Vaccinations | Phase II Arm B GM.CD40L.CCL21 Vaccinations
Serious Adverse Events (participants affected / at risk) | 1/3 | 14/37 | 7/33
Other Adverse Events (participants affected / at risk) | 3/3 | 35/37 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I GM.CD40L.CCL21 Vaccinations (N=3) | Phase II Arm A GM.CD40L Vaccinations (N=37) | Phase II Arm B GM.CD40L.CCL21 Vaccinations (N=33)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (2)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Death NOS (General disorders) | 0 (0) | 0 (0) | 5 (5)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gallbladder infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I GM.CD40L.CCL21 Vaccinations (N=3) | Phase II Arm A GM.CD40L Vaccinations (N=37) | Phase II Arm B GM.CD40L.CCL21 Vaccinations (N=33)
Injection site reaction (General disorders) | 1 (2) | 19 (39) | 21 (45)
Fatigue (General disorders) | 2 (3) | 19 (21) | 15 (18)
Edema limbs (General disorders) | 0 (0) | 5 (5) | 4 (4)
Pain (General disorders) | 0 (0) | 2 (2) | 7 (8)
Fever (General disorders) | 1 (1) | 3 (3) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 2 (3) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 3 (3) | 1 (1)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other (General disorders) | 0 (0) | 2 (4) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 11 (14) | 13 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 10 (10) | 13 (14)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 6 (8) | 11 (11)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 7 (8) | 4 (6)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 4 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 1 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 2 (2)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 3 (6) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 9 (10) | 7 (7)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (8) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 8 (9)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (5) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (7)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth development disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 6 (10) | 6 (8)
Investigations - Other (Investigations) | 0 (0) | 3 (4) | 9 (13)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (6) | 3 (6)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 3 (4)
Weight loss (Investigations) | 1 (1) | 2 (2) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (3) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 7 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 5 (6)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 5 (6)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 9 (12) | 7 (10)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Spleen disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 5 (5) | 4 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0)
Nervous system disorders - Other (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 2 (2) | 2 (3)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Papulopustular rash (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular disorders - Other (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (5) | 4 (4)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 2 (3)
Premature menopause (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes